CLINICAL TRIAL: NCT01162434
Title: Volumetric Brain MRI (Magnetic Resonance Imaging) Comparison of Patients With Treatment Resistant Depression (TRD) Undergoing Deep Brain Stimulation (DBS) With Age, Sex and Education Matched Healthy Controls
Brief Title: Brain MRI (Magnetic Resonance Imaging) Scans of Patients With Treatment Resistant Depression (TRD) and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Collaborators: North Bristol NHS Trust (Other)
Responsible Party: Dr. Birgit Whitman, University of Bristol
Other Study IDs: UoB1112; 10/H0102/15 (Other: Southmead REC)
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2011-08

CONDITIONS: Mental Disorders
Keywords: Treatment resistant depression; Deep brain stimulation; Brain volumetric analysis
MeSH Terms: conditions — Mental Disorders; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Up to 8 patients who have received Deep Brain Stimulation for Treatment Resistant Depression at Frenchay Hospital (UK) will be recruited.
- Healthy volunteers: Up to 16 healthy volunteers, matched to the DBS patients on age, sex, handedness, and education, will be recruited.

SUMMARY:
Treatment resistant depression (TRD) is a major health concern, with 10% of patients with major depressive disorder not responding to conventional treatments. The investigators propose to compare the MRI (magnetic resonance imaging) brain scans of patients with TRD, which were collected during surgical planning for deep brain stimulation, with age, sex, handedness and education-matched healthy volunteer controls, to investigate anatomical differences, specifically the volume of certain brain structures.

DETAILED DESCRIPTION:
All the patients treated at Frenchay Hospital, UK, with deep brain stimulation (DBS) for treatment resistant depression (TRD) will be given a Patient Information Sheet, and asked if they would like to participate in this research related to their condition. If they indicate they would like to participate, patients will be asked to sign a separate informed consent form (ICF) to give permission for their previously collected MRI scan to be used for this new research purpose. Information on handedness of the patients has not been previously collected, so patients will be given a short questionnaire to determine their handedness. The patients will not be required to perform any further tasks.

For each patient that agrees to participate in the study, two healthy matched control participants will be recruited. Participants will be recruited from an existing volunteer database and by local advertisements.

Respondents interested in participating will be given a letter of invite and a participant information sheet. They will be asked several basic questions including contact details, health status, age, sex, handedness, highest qualification achieved, and scanning requirements in order to assess their basic suitability for the study. If suitable, participants will be invited to attend a screening visit. Here, the informed consent form will be signed, then their medical history will be taken, and they will be given a MINI neuropsychiatric evaluation to assess their physical and mental status. Females who have the possibility of being pregnant will be asked to provide a urine sample to check they are not pregnant, and will be required to use adequate contraception until after their scan.

If suitable, participants will complete two computerised tests of mood. Then they will have a scan date booked at Frenchay hospital. At the scanning visit, participants will be assessed for any changes in health since their screening visit, and then will complete an MRI scan. The same scanner with the same sequences will be used for the healthy controls that were used for the patients. Two sequences will be collected: a coronal T1 FFE (fast field echo) volume acquisition and an axial high resolution T2 limited volume acquisition where 16 slices are collected with 8 above the ACPC (anterior commissure posterior commissure) plane and 8 below. These sequences match the sequences that our DBS patients have had and will allow both automated anatomical quantitative analysis (using Statistical Parametric Mapping version 5 (SPM5)) and quantitative description of other MRI signals such as white matter bright spots. Participants will receive no payment, but can have a printout of their scan if they wish.

The scans will then be analysed and compared to the patient scans.

ELIGIBILITY:
Inclusion Criteria:

* Up to 12 females and 4 males, sex, handedness and age (±5 years) matched for the DBS patients.

Exclusion Criteria:

* Current or past psychiatric disorder as assessed with MINI and clinical interview.
* Significant head injury.
* Standard MRI risk criteria (metallic clips or pins in body, pacemaker, aneurysm clips, pregnancy, possibility of metal in eyes including history of traumatic eye injury, shrapnel or bullet injuries).
* Inability to lie in the scanner for whatever reason (e.g. claustrophobia).
* Current acute medical illness.
* Started on new medicines in the last two months that the investigator feels may interfere with the study.
* Any medical condition that in the principle investigator's opinion is not matched in the DBS sample (e.g. epilepsy, diabetes, cardiac/hepatic/renal failure but not hypertension).
* The investigator feels that the volunteer is unsuitable for the research protocol, or unable or unwilling to comply with study procedures.

Ages: 26 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have received Deep Brain Stimulation (DBS) for Treatment Resistant Depression at Frenchay Hospital, UK., and healthy volunteers who are matched to the DBS patients, sampled from the local area.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Region of interest analysis | 6 months
  Comparison of RoI volumes of specific brain structures between patients with TRD undergoing deep brain stimulation (DBS) and healthy volunteers. Specific brain regions are: hippocampus, orbitofrontal cortex and subgenual cingulate, amygdala, dorsal anterior cingulate cortex, and dorsomedial prefrontal cortex.
Whole brain analysis | 6 months
  Whole brain MRI volumetric comparison between TRD patients undergoing DBS and healthy volunteers.
Comparison of abnormalities | 6 months
  Comparison of other potential abnormalities e.g. areas of hyperintensity in white matter in specific brain volumes between patients with TRD undergoing DBS and healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Malizia, MD, Principal Investigator — University of Bristol
Locations (1):
- Bristol Royal Infirmary, Bristol, United Kingdom